CLINICAL TRIAL: NCT06123403
Title: Evaluation of High Dose Methotrexate Toxicity in Correlation With Blood Methotrexate Level and the Role of Cystatin C in Prediction of Acute Kidney Injury in Pediatric Malignancies
Brief Title: Evaluation of High Dose Methotrexate Toxicity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hosam Hasan Khalaf, assistant lecturer, Sohag University
Other Study IDs: HD- methotrexate toxicity
Record Dates: First submitted 2023-10-27; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Methotrexate Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: blood methotrexate level and Cystatin C level — blood methotrexate level and Cystatin C level

SUMMARY:
This study aims to:

1. Evaluation of high dose methotrexate related toxicities among children admitted to Sohag Oncology Centre.
2. Role of methotrexate blood level in prediction of high dose methotrexate related toxicities.
3. Role of Cystatin C as a predictor for acute kidney injury in high dose methotrexate related toxicities.
4. Factors affecting outcome of high dose methotrexate related toxicities.

DETAILED DESCRIPTION:
It is a prospective observational study will be carried out on children receiving high dose methotrexate in Sohag Oncology Centre with one-year observation starting from January 2024.

All children receiving high dose methotrexate in Sohag Oncology Centre and fulfill the study inclusion criteria with one-year observation starting from January 2024. Informed consent will be taken from the parents/guardians.

A Prepared sheet to collect data related to this study that include:

1. Socio-demographic data: e.g. age, sex, residence in addition to dose of MTX and tumor type.
2. General and systemic manifestations: gastrointestinal manifestations, neurological manifestations, respiratory and hematological manifestations.
3. Investigations: blood samples will be collected for CBC, Urea, Creatinine, ALT, AST, Methotrexate level and Cystatin C.
4. Treatment lines: fluid, folinic acid, alkalinization of urine, blood elements, hemodialysis and colony stimulating factors.
5. Outcome: complete recovery, residual effects, complications or death.

ELIGIBILITY:
Inclusion Criteria:

* Children admitted to Sohag Oncology Centre, age from 1 to 18 years
* receive high dose methotrexate therapy equal to or more than 1 gm/m2 surface area.

Exclusion Criteria:

* WBCs less than 1000 / microliter
* Platelet count less than 50000 / microliter
* Renal affection
* Hepatic affection
* Respiratory affection
* Diabetes mellitus
* Cardiovascular disease

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children admitted to Sohag Oncology Centre, age from 1 to 18 years and receive high dose methotrexate therapy equal to or more than 1 gm/m2 surface area.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Role of methotrexate blood level in prediction of methotrexate related toxicities | baseline
  Venous blood will be collected under complete aseptic condition about 5 milliliters to measure serum methotrexate level using drug analyzer then the level of methotrexate will be used as apredictor to identify high dose methotrexate related toxicities in pediatric malignancies We will see if the test could predict the occurrence of toxicities before it happens or not
Role of Cystatin C in prediction of acute kidney injury | Baseline
  Venous samples will be collected about 3 milliliters under complete aseptic condition then centrifuged then the level of Cystatin C will be measured and will be used as abiomarker to detect acute kidney injury associated with high dose methotrexate related toxicities We will see if the test could predict occurrence of acute kidney injury before it happens or not

CONTACTS AND LOCATIONS:
Overall Officials: Maha A Helal, Professor, Study Director — Sohag University

REFERENCES:
- [Background] Barreto JN, McClanahan AL, Rule AD, Thompson CA, Frazee E. Incorporating Cystatin C to Predict Methotrexate Elimination in Patients with CNS Lymphoma and Suspicious Renal Function. Case Rep Hematol. 2018 Mar 26;2018:7169897. doi: 10.1155/2018/7169897. eCollection 2018. PMID 29780646
- [Background] Bebarta VS, Hensley MD, Borys DJ. Acute methotrexate ingestions in adults: a report of serious clinical effects and treatments. J Toxicol. 2014;2014:214574. doi: 10.1155/2014/214574. Epub 2014 Apr 16. PMID 24829573
- [Background] Bello AE, Perkins EL, Jay R, Efthimiou P. Recommendations for optimizing methotrexate treatment for patients with rheumatoid arthritis. Open Access Rheumatol. 2017 Mar 31;9:67-79. doi: 10.2147/OARRR.S131668. eCollection 2017. PMID 28435338
- [Background] Li X, Sui Z, Jing F, Xu W, Li X, Guo Q, Sun S, Bi X. Identifying risk factors for high-dose methotrexate-induced toxicities in children with acute lymphoblastic leukemia. Cancer Manag Res. 2019 Jul 5;11:6265-6274. doi: 10.2147/CMAR.S207959. eCollection 2019. PMID 31308758